CLINICAL TRIAL: NCT00733746
Title: A Phase II Study of Preoperative Gemcitabine and Erlotinib Plus Pancreatectomy and Postoperative Gemcitabine and Erlotinib for Patients With Operable Pancreatic Adenocarcinoma
Brief Title: Gemcitabine and Erlotinib Before and After Surgery in Treating Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); OSI Pharmaceuticals (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z5041; ACOSOG-Z5041; U10CA076001 (NIH); NCI-2009-00348 (Other: NCI Clinical Trial Reporting Office); CDR0000609871 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage I pancreatic cancer; stage II pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant therapy + Surgery + Adjuvant therapy (Experimental): As part of neoadjuvant therapy, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 29, 36, and 43 and oral erlotinib hydrochloride once daily on days 1-43 in the absence of disease progression or unacceptable toxicity. Within 3-6 weeks after completion of neoadjuvant therapy, patients undergo pancreaticoduodenectomy and patients receive gemcitabine hydrochloride and erlotinib hydrochloride as in neoadjuvant therapy within 5-10 weeks post surgery.
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: erlotinib hydrochloride — oral administration
Drug: gemcitabine hydrochloride — Intravenous administration
Procedure: therapeutic conventional surgery

SUMMARY:
PURPOSE: This phase II trial is studying how well gemcitabine and erlotinib work when given before and after surgery in treating patients with pancreatic cancer that can be removed by surgery. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine and erlotinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these drugs after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
This is a single arm, non-randomized phase II study. Eligible, fully registered patients will receive preoperative chemotherapy consisting of gemcitabine plus erlotinib. Preoperative chemotherapy will be followed by exploratory laparotomy and pancreaticoduodenectomy. Patients will then receive postoperative chemotherapy consisting of gemcitabine plus erlotinib. Up to 123 patients will be accrued to this study, with the expectation that 78 patients will remain fully eligible and evaluable for the primary endpoint. The primary and secondary objectives for the study are listed below.

Primary Objective:

To estimate the proportion of patients alive at two years from the date of registration

Secondary Objectives:

1. To determine the resection rate (defined as the fraction of patients who proceed to planned surgery with removal of primary tumor [R0/R1]) following induction treatment with gemcitabine plus erlotinib
2. To estimate the time to disease progression/relapse
3. To evaluate the rate of R0, R1, and R2 resections (defined as per the 6th edition of the AJCC Cancer Staging Manual) in patients treated with preoperative gemcitabine plus erlotinib chemotherapy
4. To evaluate the toxicity profile of preoperative gemcitabine plus erlotinib and the feasibility of postoperative gemcitabine plus erlotinib
5. To evaluate response rates to preoperative chemotherapy for patients treated with preoperative gemcitabine and erlotinib
6. To identify molecular predictors of pancreatic cancer response to gemcitabine combined with erlotinib
7. To identify genetic profiles of pancreatic adenocarcinoma that may be associated with response to neoadjuvant therapy

After completion of postoperative chemotherapy treatment, patients are followed every 3 months for 2 years and then every 6 months for 2 years.

ELIGIBILITY:
Eligibility Criteria:

1. Cytologic or histologic proof of adenocarcinoma of the pancreatic head or uncinate process.

   NOTE: Patients with tumors of the pancreatic neck, body or tail are not eligible. Patients with evidence of neuroendocrine tumors, duodenal adenocarcinoma, or ampullary adenocarcinoma are not eligible.
2. Localized, potentially resectable tumors as defined below. All patients must be staged with a chest X-ray or CT, and abdominal CT (contrast-enhanced, helical thin-cut) or MRI. Radiological resectability is defined by the following criteria on abdominal imaging:

   * No evidence of tumor extension to the celiac axis, hepatic artery, or superior mesenteric artery
   * No evidence of tumor encasement or occlusion of the superior mesenteric vein (SMV) or the SMV/portal vein confluence
   * No evidence of visceral or peritoneal metastases

   NOTE: Patients with borderline resectable or marginally resectable pancreatic cancer are not eligible. Patients must meet all objective imaging criteria outlined above.
3. ≥ 18 years of age
4. ECOG/Zubrod performance status of 0 or 1
5. Baseline weight loss ≤ 15% of premorbid weight
6. Patient must have adequate hematologic, renal, and hepatic function as defined by:

   * WBC ≥ 2,000 cells/mm³
   * ANC ≥ 1,500 cells/mm³
   * Platelets ≥ 100,000 cells/mm³
   * Serum bilirubin ≤ 2.5 mg/dL
   * Serum creatinine ≤ 1.5 mg/dL or a calculated creatinine clearance of ≥ 50 ml/min (24 hour urine collection)
   * ALT < 2.5 times upper limit of normal (ULN)
   * AST < 2.5 times ULN
   * Albumin ≥ 3.2 g/dl
7. No history of the following:

   * Prior EGFR targeted therapy or therapy for pancreatic cancer
   * Active infection requiring intravenous antibiotics at the time of registration
8. Non-pregnant and non-breast feeding. Female participants of child bearing potential must have a negative urine or serum pregnancy test prior to registration. Perimenopausal participants must be amenorrheic ≥ 12 months to be considered not of childbearing potential. All patients of reproductive potential must agree to use an effective method of birth control while receiving study therapy.
9. No prior malignancy within 5 years of registration (Exceptions: non-melanoma skin cancer, in-situ cancers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2019-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W.T. Pisters, MD, Study Chair — M.D. Anderson Cancer Center
Locations (24):
- United States (23):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Surgical Oncology Associates, Newport News, Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
- Princess Margaret Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 123 patients enrolled to this study. 4 patients cancelled prior to treatment and were not included in any analysis.
Groups:
- Neoadjuvant Therapy + Surgery + Adjuvant Therapy: Neoadjuvant Therapy:
  As part of neoadjuvant therapy, patients receive 1000 mg/m2 gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 15, 29, 36, and 43 and 100 mg oral erlotinib hydrochloride once daily on days 1-43 in the absence of disease progression or unacceptable toxicity.
  Surgery:
  Within 3-6 weeks after completion of neoadjuvant therapy, patients are reevaluated for eligibility for pancreaticoduodenectomy.
  Adjuvant Therapy:
  Patients that receive pancreaticoduodenectomy according to protocol are given 1000 mg/m2 gemcitabine hydrochloride IV on days 1, 8, 15, 29, 36, and 43 and 100 mg erlotinib hydrochloride as in neoadjuvant therapy within 5-10 weeks post-surgery.
Period: Overall Study
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Started | 119
Completed | 114
Not Completed | 5
Not completed — Ineligible | 5

BASELINE CHARACTERISTICS:
Population: All patients that started protocol treatment were included in this analysis.
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Number analyzed (Participants) | 119
Age, Continuous [Median (Full Range); unit: years] | 66 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 61
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 19
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 2 Years
Description: The primary endpoint of this trial is 2-year overall survival, which will be evaluated as the proportion of treatment successes. A treatment success is defined to be an evaluable patient who is alive at two years from the date of registration.
Time Frame: At 2 years post-registration
Population: All patients meeting the eligibility criteria who completed neoadjuvant therapy and underwent protocol surgery with R0 or R1 resection were evaluated for the primary endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Number analyzed (Participants) | 74
proportion of patients | 0.54 [0.42 to 0.66]

2. Secondary Outcome: Resection Rate
Description: The resection rate is defined as the fraction of patients that proceed to planned surgery with removal of primary tumor (R0/R1) following neoadjuvant treatment with gemcitabine plus erlotinib.The resection rate will be estimated by the binomial point estimate, i.e. as the number of patients that undergo the planned surgery with removal of the primary tumor following neoadjuvant treatment with gemcitabine plus erlotinib divided by the number of evaluable patients. This quantity will also be estimated with a 95% binomial confidence interval.
  Curative resection (R0) is defined as macroscopically and microscopically complete resection (with microscopic surgical margin assessment according to AJCC Staging Principles).
  An R1 resection is defined as macroscopically complete tumor removal with any positive microscopic surgical margin (bile duct, pancreatic parenchyma, or SMA margins).
Time Frame: Up to 4 years postoperative chemotherapy treatment
Population: All patients that completed neoadjuvant treatment and were eligible for surgery were included in this endpoint.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: proportion of patients
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Number analyzed (Participants) | 97
proportion of patients | 0.76 [0.67 to 0.84]

3. Secondary Outcome: Relapse/Progression-free Survival
Description: Relapse/progression-free survival is defined as the time from date of registration to the date of documentation of disease recurrence/progression. If a patient dies without documentation of disease recurrence/progression, the patient will be considered to have had disease recurrence/progression at the time of their death unless there is sufficient documented evidence to conclude no recurrence/progression occurred prior to death. If a patient is declared to be a major treatment violation, the patient will be censored on the date the treatment violation occurred. If a patient is lost to follow-up, s/he will be censored at the data of last contact. The distribution of disease-free survival will be estimated using the method of Kaplan and Meier.
Time Frame: At 2 years post-registration
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Number analyzed (Participants) | 74
months | 11.9 [10.8 to 17.5]

4. Secondary Outcome: Number of Participants Experiencing Grade 3 or Higher Adverse Events as Graded by the NCI's Common Toxicity Criteria for Adverse Events
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns. These patterns will be summarized with descriptive statistics. The number of patients reporting grade 3 or higher adverse events as graded by the NCI's Common Toxicity Criteria (CTCAE) Version 4 are reported here. A complete list of all reported adverse events is reported in the Adverse Events section of this report.
Time Frame: Up to 4 years postoperative chemotherapy treatment
Population: All patients that started protocol treatment and were assessed for adverse events were included in this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Number analyzed (Participants) | 119
Participants
  Grade 3+ Adverse Event | 27
  Grade 4+ Adverse Event | 2

5. Secondary Outcome: Response Rate
Description: The response rates to preoperative chemotherapy for patients treated with preoperative gemcitabine and erlotinib and rates of accurate pathologic assessment of the resected tumor specimen according to College of American Pathology guidelines will be estimated with a binomial point estimate and corresponding 95% confidence intervals.
Time Frame: Up to 4 years postoperative chemotherapy treatment
Population: All patients that completed neoadjuvant treatment and were eligible for protocol surgery were included in this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Number analyzed (Participants) | 97
proportion of patients | 0.06 [0.02 to 0.13]

ADVERSE EVENTS:
Arm/Group | Neoadjuvant Therapy + Surgery + Adjuvant Therapy
Serious Adverse Events (participants affected / at risk) | 37/119
Other Adverse Events (participants affected / at risk) | 118/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Therapy + Surgery + Adjuvant Therapy (N=119)
Hemoglobin decreased (Blood and lymphatic system disorders) | 5 (5)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 4 (5)
Localized edema (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 6 (6)
Endocarditis infective (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (8)
Amylase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 9 (9)
Bilirubin increased (Investigations) | 6 (6)
Creatinine increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Therapy + Surgery + Adjuvant Therapy (N=119)
Blood disorder (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 96 (146)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Endocrine disorder (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3)
Conjunctival disorder (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 7 (10)
Eye disorder (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 27 (30)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 22 (22)
Diarrhea (Gastrointestinal disorders) | 58 (74)
Dry mouth (Gastrointestinal disorders) | 21 (25)
Dyspepsia (Gastrointestinal disorders) | 39 (43)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 10 (11)
Gastrointestinal disorder (Gastrointestinal disorders) | 5 (5)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 66 (79)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 34 (35)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 10 (11)
Edema limbs (General disorders) | 16 (17)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 90 (125)
Fever (General disorders) | 21 (22)
Flu-like symptoms (General disorders) | 2 (2)
General symptom (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 11 (12)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Otitis externa (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative gastrointestinal injury - Oral cavity NOS (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 83 (114)
Alkaline phosphatase increased (Investigations) | 24 (28)
Amylase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 76 (108)
Bilirubin increased (Investigations) | 46 (49)
Coagulopathy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 10 (10)
Gamma-glutamyltransferase increased (Investigations) | 6 (6)
INR increased (Investigations) | 4 (4)
Laboratory test abnormal (Investigations) | 6 (11)
Leukocyte count decreased (Investigations) | 76 (109)
Lipase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 18 (23)
Neutrophil count decreased (Investigations) | 46 (59)
Pancreatic enzymes decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 82 (119)
Serum cholesterol increased (Investigations) | 2 (2)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 14 (14)
Anorexia (Metabolism and nutrition disorders) | 30 (32)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 42 (60)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 4 (5)
Serum albumin decreased (Metabolism and nutrition disorders) | 28 (31)
Serum calcium decreased (Metabolism and nutrition disorders) | 15 (17)
Serum glucose decreased (Metabolism and nutrition disorders) | 5 (6)
Serum magnesium decreased (Metabolism and nutrition disorders) | 5 (6)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 8 (8)
Serum potassium decreased (Metabolism and nutrition disorders) | 23 (28)
Serum potassium increased (Metabolism and nutrition disorders) | 5 (5)
Serum sodium decreased (Metabolism and nutrition disorders) | 16 (21)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (5)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 16 (18)
Memory impairment (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6)
Taste alteration (Nervous system disorders) | 32 (39)
Tremor (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 10 (11)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 11 (12)
Urinary frequency (Renal and urinary disorders) | 5 (5)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (26)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 30 (39)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 35 (42)
Rash acneiform (Skin and subcutaneous tissue disorders) | 79 (108)
Rash desquamating (Skin and subcutaneous tissue disorders) | 38 (43)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (6)
Sweating (Skin and subcutaneous tissue disorders) | 3 (4)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 11 (12)
Hypotension (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less